CLINICAL TRIAL: NCT02527564
Title: A Double-blind, Randomized, Placebo-controlled Trial of Adjunctive Suvorexant for Treatment-resistant Insomnia in Patients With Bipolar Disorder
Brief Title: Efficacy of Suvorexant to Treat Insomnia Related to Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Po W Wang, Clinical Professor, Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 53208
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Insomnia; Bipolar Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Bipolar Disorder | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suvorexant (Experimental): 50% of enrolled participants will be randomly assigned to receive double-blind suvorexant for one week, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the last 4 nights.
  Following the one-week double-blind, placebo-controlled phase, 100% of participants will receive open-label suvorexant for 3 months, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the remainder of 3 months.
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): 50% of enrolled participants will be randomly assigned to receive double-blind placebo pill for one week, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the last 4 nights.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant
  Other Names: Belsomra
  Arms: Suvorexant
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of suvorexant, added to existing medications, for treatment-resistant insomnia in individuals with bipolar disorder. The investigators hypothesize that participants receiving suvorexant for one week will experience significantly greater improvement in sleep duration compared to participants receiving placebo.

DETAILED DESCRIPTION:
Participants will be randomized to receive double-blind suvorexant or placebo for one week, after which all participants will receive open treatment with suvorexant for three months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatients meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for bipolar I disorder (296.70), bipolar II disorder (296.89), or bipolar disorder not otherwise specified (296.80), with concurrent insomnia related to bipolar disorder (307.42).
2. Currently taking ≥ 1 prescription psychotropic medication (hypnotic agents, anxiolytics, atypical antipsychotics, mood stabilizers, and/or antidepressants) for management of bipolar disorder.
3. Subjective total sleep time (sTST) < 6 hours on ≥ 1 night during the prior week.

Exclusion Criteria:

1. Current hypo/manic symptoms, as evidenced by the Young Mania Rating Scale (YMRS) total score ≥ 12.
2. Current (past 6 months) alcohol or substance use disorder.
3. Current psychosis.
4. Patients who are actively suicidal or evaluated as being a high suicide risk.
5. Women who are currently pregnant or breastfeeding.
6. Clinically significant abnormalities on baseline laboratory tests (comprehensive metabolic panel, fasting lipid panel, Complete Blood Count (CBC) with differential, thyroid stimulating hormone).
7. Presence of any unstable and/or potentially confounding neurological and/or medical disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-09; Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Po Wang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 61 participants consented, 48 participants were randomized to a study arm.
Groups:
- Suvorexant (Double-blind): Participants receive double-blind suvorexant for one week, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the last 4 nights.
- Placebo (Double-blind): Participants receive double-blind placebo to match suvorexant for one week.
- Suvorexant (Open-label): Participants receive open-label suvorexant for 3 months, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the remainder of 3 months.
Period: Double-blind Phase (1 Week)
Arm/Group | Suvorexant (Double-blind) | Placebo (Double-blind) | Suvorexant (Open-label)
Started | 23 | 25 | 0
Received Allocated Intervention | 19 | 17 | 0
Completed | 22 | 24 | 0
Not Completed | 1 | 1 | 0
Period: Open-label Phase (3 Months)
Arm/Group | Suvorexant (Double-blind) | Placebo (Double-blind) | Suvorexant (Open-label)
Started | 0 | 0 | 46 (Participants who continued after the double-blind phase are represented in the Suvorexant (open-label) group.)
Completed | 0 | 0 | 26
Not Completed | 0 | 0 | 20

BASELINE CHARACTERISTICS:
Population: Participants who received the allocated intervention are included in the analysis
Groups:
- Suvorexant: Participants receive double-blind suvorexant for one week, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the last 4 nights. Following the double-blind phase, participants receive open-label suvorexant for 3 months, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the remainder of 3 months.
- Placebo: Participants receive double-blind placebo to match suvorexant for one week. Following the double-blind phase, participants receive open-label suvorexant for 3 months, dosed at 10mg every bedtime for the first 3 nights, then increased to 20mg every bedtime for the remainder of 3 months.
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.84 (14.792) | 44.53 (14.841) | 48.92 (15.197)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 1 | 2 | 3
  Hispanic | 0 | 2 | 2
  White | 12 | 9 | 21
  Multi/Other | 5 | 3 | 8
  Unknown | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Total Sleep Time - Acute
Description: Measured by self-report electronic sleep diary. Change is calculated as week 1 value minus week 0 value.
Time Frame: baseline and week 1 of double-blind, placebo-controlled phase
Population: Participants who received the allocated intervention and with data at all time points are included in the analysis. This outcome was assessed in the double-blind groups only.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant (Double-blind) | Placebo (Double-blind)
Number analyzed (Participants) | 14 | 10
hours
  week 0 | 7.04 (1.16) | 7.03 (0.55)
  week 1 | 7.53 (1.43) | 7.20 (0.68)
  change at week 1 | 0.49 (1.03) | 0.17 (0.90)
Statistical Analysis 1: Comparison: Suvorexant (Double-blind); Within group change at week 1 - suvorexant (double-blind); Test type: Other; p = 0.10, Paired 2-sided t-test — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Placebo (Double-blind); Within group change at week 1- placebo (double-blind) group; Test type: Other; p = 0.57, Paired 2-sided t-test — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 3: Comparison: Suvorexant (Double-blind) vs Placebo (Double-blind); Between group change at week 1; Test type: Other; p = 0.44, Unpaired 2-sided t-test — A p-value of <0.05 would be considered statistically significant

2. Secondary Outcome: Change in Objective Total Sleep Time - Acute
Description: Measured by actigraphy. Change is calculated as week 1 value minus week 0 value.
Time Frame: baseline and week 1 of double-blind, placebo-controlled phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant (Double-blind) | Placebo (Double-blind)
Number analyzed (Participants) | 14 | 10
hours
  week 0 | 6.46 (2.06) | 9.50 (4.64)
  week 1 | 7.20 (2.60) | 10.10 (4.10)
  change at week 1 | 0.74 (1.17) | 0.61 (3.15)
Statistical Analysis 1: Comparison: Suvorexant (Double-blind); Within group change at week 1 - suvorexant (double-blind); Test type: Other; p = 0.035, Paired 2-sided t-test — A p-value of <0.05 would be considered significantly significant
Statistical Analysis 2: Comparison: Placebo (Double-blind); Within group change at week 1- placebo (double-blind) group; Test type: Other; p = 0.55, Paired 2-sided t-test; A p-value of <0.05 would be considered statistically significant
Statistical Analysis 3: Comparison: Suvorexant (Double-blind) vs Placebo (Double-blind); Between group change at week 1; Test type: Other; p = 0.89, Paired 2-sided t-test — A p-value of <0.05 would be considered statistically significant

3. Secondary Outcome: Subjective Total Sleep Time - Subchronic
Description: Measured by self-report electronic sleep diary. Change is calculated as the month 3 value minus the week 1 value
Time Frame: week 1 and month 3 of open treatment phase
Population: Participants who received the allocated intervention and with data at all time points are included in the analysis. Month 3 data were collected using last observation carried forward method (LOCF). This outcome was assessed in the open-label group only.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant (Open-label)
Number analyzed (Participants) | 24
hours
  week 1 | 7.24 (1.32)
  month 3 | 7.25 (1.56)
  change at month 3 | 0.01 (1.29)
Statistical Analysis 1: Comparison: Suvorexant (Open-label); Within group change at month 3 - suvorexant (open-label); Test type: Other; p = 0.97, Paired 2-sided t-test — A p-value of <0.05 would be considered significantly significant

4. Secondary Outcome: Change in Objective Total Sleep Time - Subchronic
Description: Measured by actigraphy. Change is measured as the month 3 value minus the week 1 value.
Time Frame: week 1 and month 3 of open treatment phase
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant (Open-label)
Number analyzed (Participants) | 24
hours
  week 1 | 8.69 (3.44)
  month 3 | 9.58 (4.56)
  change at month 3 | 0.88 (3.82)
Statistical Analysis 1: Comparison: Suvorexant (Open-label); Within group change at month 3 - suvorexant (open-label); Test type: Other; p = 0.28, Paired 2-sided t-test — A p-value of <0.05 would be considered significantly significant

ADVERSE EVENTS:
Time Frame: 1 week in the double-blind phase, and 3 months in the open-label phase
Arm/Group | Suvorexant (Double-blind) | Placebo (Double-blind) | Suvorexant (Open-label)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/25 | 0/46
Other Adverse Events (participants affected / at risk) | 1/23 | 1/25 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (Double-blind) (N=23) | Placebo (Double-blind) (N=25) | Suvorexant (Open-label) (N=46)
Breast Drainage (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (Double-blind) (N=23) | Placebo (Double-blind) (N=25) | Suvorexant (Open-label) (N=46)
Hypersomnolence (Psychiatric disorders) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT02527564/Prot_SAP_000.pdf